CLINICAL TRIAL: NCT03642756
Title: Effects of Different Intra-arterial Catheter Size on the Frequency of Optimal Dynamic Response in Radial Arterial Waveform
Brief Title: Effects of Different Intra-arterial Catheter Size on Frequency of Optimal Dynamic Response in Radial Arterial Waveform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: catheter size
Record Dates: First submitted 2018-07-27; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Catheters

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 gauge (Placebo Comparator)
  Interventions: Device: different intra-arterial catheter size
- 22 gauge (Active Comparator)
  Interventions: Device: different intra-arterial catheter size
- 24 gauge (Active Comparator)
  Interventions: Device: different intra-arterial catheter size

INTERVENTIONS:
Device: different intra-arterial catheter size — in placebo group, patients were cannulated with 20 gauge intra-arterial catheter. In experiment groups, patients were cannulated with 22 gauge or 24 gauge intra-arterial catheter.

SUMMARY:
The aim of this study is to compare the effects of different intra-arterial catheter size on the frequency of optimal dynamic response in radial arterial waveform.

ELIGIBILITY:
Inclusion Criteria:

* patients who were scheduled for elective neurosurgery under general anesthesia
* patients with age of 20-79 and ASA class I-III
* patients who are needed to establish invasive arterial pressure monitoring

Exclusion Criteria:

* patients who refuted to be involved in the study
* patients with age of <20 or >80
* patients who had both arm saved
* patients who had a previous history of surgery on radial artery

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of adequately damped arterial waveform | 1 minute after cannulation
  The accuracy of arterial blood pressure waveform is depedent on damping coefficient (DC) and natural frequency (NF). The extent to which a monitoring system is damped is expressed by the DC, while the frequency of oscillation that a monitoring system resonates at is known as the NF. The NF and DC are required to be within certain rages for accurate blood pressure monitoring, and they can be affected by different arterial catheter size. Adequately damped arterial waveform can be defined as NF and DC being within certain ranges. For example, waveforms with DC of 0.5 at a NF of 15Hz can be regarded as adequately damped arterial waveform. However, if waveforms have DC of 0.1 at a NF of 15Hz, these can be regarded as not having optimal dynamic response. (There is a reference figure explaining these factors in detail in a previous article. Gardner RM: Direct blood pressure measurement--dynamic response requirements. Anesthesiology 1981; 54:227-3)

SECONDARY OUTCOMES:
The difference of mean blood pressure between invasive blood pressure and non-invasive blood pressure | 1 minute after cannulation
  At 1 minute after cannulating radial artery, we will obtain information about the mean blood pressure measured in both invasive blood pressure and non-invasive blood pressure. Invasive blood pressure will be measured from radial artery cannulation, and non-invasive blood pressure will be measured by blood pressure cuff at Rt. upper arm. Thereafter, the difference of mean blood pressure between two values will be used for data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh H, Choe SH, Kim YJ, Yoon HK, Lee HC, Park HP. Intraarterial catheter diameter and dynamic response of arterial pressure monitoring system: a randomized controlled trial. J Clin Monit Comput. 2022 Apr;36(2):387-395. doi: 10.1007/s10877-021-00663-7. Epub 2021 Feb 1. PMID 33527182